CLINICAL TRIAL: NCT01724502
Title: PGC-1 and Mitochondrial Dysfunction in Diabetes, Aims 4 & 5
Brief Title: Mitochondrial Dysfunction in Diabetes
Acronym: PGC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lawrence Mandarino, Ph.D., Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-006065 Aim 4; R01DK066483 (NIH)
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes; Obese
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Obese Non-Diabetic Subjects (Experimental): All subjects on this arm will undergo exercise and muscle biopsies.
  Interventions: Behavioral: Exercise and muscle biopsies
- Type 2 Diabetic Subjects (Experimental): All subjects on this arm will undergo exercise and muscle biopsies.
  Interventions: Behavioral: Exercise and muscle biopsies
- Healthy Control Subjects (Experimental): All subjects on this arm will undergo exercise and muscle biopsies.
  Interventions: Behavioral: Exercise and muscle biopsies

INTERVENTIONS:
Behavioral: Exercise and muscle biopsies — Subjects will undergo a euglycemic clamp, VO_2 max determination, exercise periods and muscle biopsies.

SUMMARY:
The purpose of this study is to determine whether insulin resistance is accompanied by "exercise resistance". Investigators will use mass spectrometry and proteomics analysis to test the hypothesis is that a bout of exercise that increases mitochondrial protein abundance in lean, healthy individuals is less effective in insulin resistant patients.

DETAILED DESCRIPTION:
The investigators' prior research has focused on defining the changes in expression of nuclear encoded mitochondrial genes that predict changes in insulin sensitivity in skeletal muscle, with the goal of defining the molecular mechanisms underlying the connection between mitochondrial dysfunction and insulin resistance in skeletal muscle.

Three groups of subjects will be studied: lean, healthy control subjects (n=12) obese non-diabetic subjects (n=12) and patients with type 2 Diabetes Mellitus (n=12) for a total of 36 subjects. Twenty subjects have completed the study at Arizona State University; the remaining 16 subjects will be accrued at the Mayo Clinic in Arizona.

Subjects will come to the Mayo Clinic 4 times. On Study Day 1 Subjects will be screened with a medical history & physical and a 75 g oral glucose tolerance test to determine if they are eligible for the study. On Study Day 2, subjects will report to the clinic after an overnight fast, undergo a euglycemic clamp (using deuterated glucose) to determine insulin sensitivity, and in addition have a muscle biopsy (basal biopsy for comparison). On Study Day 3, subjects will report to the clinic after an overnight fast, and undergo a Volume Oxygen Maximum (VO_2 max) determination. On Study Day 4, subjects will report to the clinic after an overnight fast to perform an exercise bout with muscle biopsy 30 minutes after the end of exercise. This will be followed by an overnight fast, and an additional muscle biopsy at 24 hours post exercise.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
2. Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.
3. Subjects must range in age as described in each specific protocol.
4. Subjects must have the following laboratory values:

   1. Hematocrit ≥ 35 vol%
   2. Serum creatinine ≤ 1.6 mg/dl
   3. Aspartate Aminotransferase (AST) (SGOT) < 2 times upper limit of normal
   4. Alanine Aminotransferase (ALT) (SGPT) < 2 times upper limit of normal
   5. Alkaline phosphatase < 2 times upper limit of normal
   6. Triglycerides < 150 mg/dl.
   7. Prothrombin Time (PT) 11.7 -14.3 seconds (during Intralipid/heparin infusion,PT will be determined to insure that it is < 1.5-2.0 times the normal value.)
   8. Partial thromboplastin time (PTT) 23.0-37.0 seconds.

Exclusion Criteria

1. Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for the past three months before entry into the study. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months. Subjects taking systemic glucocorticoids are excluded.
2. Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
3. Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP>180, diastolic BP>105, autonomic neuropathy, resting heart rate >100, electrolyte abnormalities.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Protein Concentration of Mitochondria | Study Day 4 (30 min after exercise) and (24 hours after exercise)
  Protein concentration will be determined from muscle biopsies by the method of Lowry. 75 micrograms of muscle lysate proteins will be separated on a 10% Sodium Dodecyl Sulfate Polyacrylamide Gel, and then visualized with Coomassie stain. The gel lane will be cut into cubes, digested with trypsin and cleaned, then protein abundance will be determined using spectral counting.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Mandarino, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States